CLINICAL TRIAL: NCT03885557
Title: Comparison Between Dynamic Oscillatory Stretch Technique and Static Stretching In Reduced Hamstring Flexibility in Healthy Population: A Single Blind Randomized Control Trial
Brief Title: Dynamic Oscillatory Stretch Technique Versus Static Stretching In Reduced Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Kanza Masood
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Hamstring Tightness
Keywords: Flexibility; Extensibility; Static stretching

STUDY DESIGN:
Who Masked: Participant
Masking Description: This was a single blind randomized control trial in which study participants were randomly allocated in 2 groups by sealed envelope methods
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I Experimental Dynamic oscillatory stretch(DOS) (Experimental): Dynamic oscillatory stretch technique (30 repetitions each of 2 seconds stretch duration in one session) was applied to DOS group.
  Interventions: Other: Group I Experimental DOS
- Group II Static Stretching(SS) Group (Active Comparator): Static stretching (2 repetitions each of 30 seconds in one session) was applied to SS group.
  Interventions: Other: group II SS group

INTERVENTIONS:
Other: Group I Experimental DOS — After the application of hot pack treatment of 7-10 minutes, dynamic oscillatory stretch(DOS) technique (30 repetitions each of 2 seconds stretch duration in one session) was applied to DOS group. An experienced orthopedic manual physical therapist provided these techniques to patients .
  Arms: Group I Experimental Dynamic oscillatory stretch(DOS)
Other: group II SS group — After the application of hot pack treatment of 7-10 minutes , Static stretching (2 repetitions each of 30 seconds in one session) was applied to SS group. An experienced orthopedic manual physical therapist provided these techniques to patients .
  Arms: Group II Static Stretching(SS) Group

SUMMARY:
This study compared the effects of dynamic oscillatory stretch technique (DOS) and static stretching (SS) technique in order to improve hamstring extensibility in healthy individuals with asymptomatic hamstring tightness. Half of study participants received DOS whereas other half received static stretching technique.

DETAILED DESCRIPTION:
This was a single blind randomized control trial conducted at District Head Quarter teaching hospital Sargodha, Sargodha institute of health sciences Sargodha, Sadiq hospital Sargodha (march 2018-June 2018). Sample size of 83 individuals was calculated through Open Epi tool version 3 with 95 % confidence interval (CI), and power 80%. 83 individuals were screened out on the basis of inclusion and exclusion criteria. Individuals of this selected population were randomly allocated as 42 individuals in Dynamic Oscillatory Stretch(DOS) group and 41 individuals in Static Stretching(SS) group by sealed envelope method.

After the application of hot pack treatment of 7-10 minutes to both groups dynamic oscillatory stretch technique (30 repetitions each of 2 seconds stretch duration in one session) was applied to DOS group and SS stretching (2 repetitions each of 30 seconds in one session) was applied to SS group.

Assessment was done at baseline, immediate post-intervention levels (immediately) and post-intervention level after 1 hour. At baseline and immediately post-intervention level there was no dropout but after 1 hour post-intervention level there were two dropouts from DOS group and 1 dropout from SS group. 40 individuals were analyzed in each DOS and SS group. Data analysis was done through Statistical Package of Social Sciences(SPSS) version 20. Normality of different variables was assessed. Shapiro-Wilk test provided the basis for normality distribution of data.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with age limit 20 to 40 years,
* Active knee extension/90-90 test positive for Screening (With AKE range less than 160 degrees),
* No known history of hip joint or knee joint disease,
* No history of recent hamstring strain.

Exclusion Criteria:

* History of sub-acute and chronic back pain of lumber region and SI joint in past 6 months,
* Neurological pathology,
* Patients with some kind of particularly specific pathology (e.g. infection, tumor, osteoporosis, lumbar spine fracture, structural deformity, inflammatory disorder).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Active Straight Leg Raise Test(ASLR) Immediate effect | 10 minutes
  Changes from baseline Active Straight Leg Raise Test(ASLR) was conducted with the participants in supine lying with both lower limbs initially extended. Then patient actively lifted the leg to be tested at hip joint while stabilizing the leg opposite to that of the testing side by using a stabilization belt. Knee on testing side was essentially sustained in full extension throughout the full testing range. Universal goniometer was used to measure range of motion available at hip joint.
  Cut off score for the SLR to indicate hamstring tightness is 80 degrees. Therefore, values of SLR below 80 degrees was considered as hamstring tightness. Assessment was done Immediate after giving intervention(10 minutes).
Active Straight Leg Raise Test(ASLR) 1 hour effects | 1 hour
  Changes from Baseline Active Straight Leg Raise Test(ASLR) was conducted with the participants in supine lying with both lower limbs initially extended. Then patient actively lifted the leg to be tested at hip joint while stabilizing the leg opposite to that of the testing side by using a stabilization belt. Knee on testing side was essentially sustained in full extension throughout the full testing range. Universal goniometer was used to measure range of motion available at hip joint.
  Cut off score for the SLR to indicate hamstring tightness is 80 degrees. Therefore, values of SLR below 80 degrees was considered as hamstring tightness. Assessment was done after 1 hour of intervention.
Active Knee Extension Test (AKE) immediate effect | 10 minutes
  Changes from Baseline Active knee extension test (AKE), is used to assess hamstring length. It was performed while the participant was in supine lying and involved leg was in 90 degree hip flexion. then participant was asked to extend the knee. For hamstring tightness cut off score AKE angle is 160°. Therefore normal individuals with angle < 160° were considered as individuals with hamstring tightness.Its reliability is 0.94.Assessment was done Immediate after giving intervention(10 minutes).
Active Knee Extension Test (AKE) 1 hour effects | 1 hour
  Changes from Baseline Active knee extension test (AKE), is used to assess hamstring length. It was performed while the participant was in supine lying and involved leg was in 90 degree hip flexion. then participant was asked to extend the knee. For hamstring tightness cut off score AKE angle is 160°. Therefore normal individuals with angle < 160° were considered as individuals with hamstring tightness.Its reliability is 0.94. Assessment was done after 1 hour of intervention.
Sit and Reach Test (SRT) Immediate effects | 10 minutes
  Changes from Baseline Sit and reach test (SRT) is most commonly employed test to measure hamstring flexibility. This tool is used to measure range of hamstring muscle at knee joint.Each participant was instructed to sits on a couch in long sitting position. participants were seated with elongated legs, with hip flexed to 90 degrees and knees were fully extended and the ankles were in relaxed plantar flexion. A measuring ruler/tape was placed,between the feet with 38 cm score was marked tangent to the sole of the feet. Subjects were asked to reach forward with hands one above the other and palms of the hands facing down, while attempting to touch fingertips to toes or as far beyond on measuring tape while keeping the knees straight. Assessment was done Immediate after giving intervention(10 minutes).
Sit and Reach Test (SRT) 1 hours effects | 1 hour
  Changes from Baseline Sit and reach test (SRT) is most commonly employed test to measure hamstring flexibility. This tool is used to measure range of hamstring muscle at knee joint.Each participant was instructed to sits on a couch in long sitting position. participants were seated with elongated legs, with hip flexed to 90 degrees and knees were fully extended and the ankles were in relaxed plantar flexion. A measuring ruler/tape was placed,between the feet with 38 cm score was marked tangent to the sole of the feet. Subjects were asked to reach forward with hands one above the other and palms of the hands facing down, while attempting to touch fingertips to toes or as far beyond on measuring tape while keeping the knees straight. Assessment was done after 1 hour of intervention.
Passive Straight Leg Raise Test(PSLR) Immediate effects | 10 minutes
  Changes from Baseline PSLR test was conducted with the participants in supine lying with both lower limbs initially extended. Then therapist lifted the leg to be tested at hip joint while stabilizing the leg opposite to that of the testing side by using a stabilization belt. Knee on testing side was essentially sustained in full extension throughout the full testing range. Universal goniometer was used to measure range of motion available at hip joint.
  Cut off score for the SLR to indicate hamstring tightness is 80 degrees. Therefore, values of SLR below 80 degrees was considered as hamstring tightness. Assessment was done Immediate after giving intervention(10 minutes).
Passive Straight Leg Raise Test(PSLR) 1 hour effects | 1 hour
  Changes from Baseline PSLR test was conducted with the participants in supine lying with both lower limbs initially extended. Then therapist lifted the leg to be tested at hip joint while stabilizing the leg opposite to that of the testing side by using a stabilization belt. Knee on testing side was essentially sustained in full extension throughout the full testing range. Universal goniometer was used to measure range of motion available at hip joint.
  Cut off score for the SLR to indicate hamstring tightness is 80 degrees. Therefore, values of SLR below 80 degrees was considered as hamstring tightness. Assessment was done after 1 hour of intervention.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) Immediate effects | 10 minutes
  Changes from Baseline Numeric pain scale (NPRS) was used to assess pain intensity. it was used to assess the tolerance ability of individuals for pain produced at the end of passive straight leg raise (PSLR) test.It ranges from 0-10. 0 means No pain and 10 means severe pain. Assessment was done after 10 minutes of intervention.
Numeric Pain Rating Scale NPRS 1 hour effects | 1 hour
  Changes from Baseline Numeric pain scale (NPRS) was used to assess pain intensity. it was used to assess the tolerance ability of individuals for pain produced at the end of passive straight leg raise (PSLR) test.It ranges from 0-10. 0 means No pain and 10 means severe pain.Assessment was done after 1 hour of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Sargodha institute of health sciences,DHQ teaching hospital Sargodha, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellote-Caballero Y, Valenza MC, Puentedura EJ, Fernandez-de-Las-Penas C, Alburquerque-Sendin F. Immediate Effects of Neurodynamic Sliding versus Muscle Stretching on Hamstring Flexibility in Subjects with Short Hamstring Syndrome. J Sports Med (Hindawi Publ Corp). 2014;2014:127471. doi: 10.1155/2014/127471. Epub 2014 Apr 15. PMID 26464889
- [Background] Youdas JW, Haeflinger KM, Kreun MK, Holloway AM, Kramer CM, Hollman JH. The efficacy of two modified proprioceptive neuromuscular facilitation stretching techniques in subjects with reduced hamstring muscle length. Physiother Theory Pract. 2010 May;26(4):240-50. doi: 10.3109/09593980903015292. PMID 20397858
- [Background] Sambandam CE, Alagesan J, Shah S. Immediate Effect of Muscle Energy Technique and Eccentric Training on Hamstring Tightness of Healthy Female Volunteers-A Comparative Study. International journal of current research and review. 2011;3(9):122-26.
- [Background] Iwasaki R, Yokoyama G, Kawabata S, Suzuki T. Lumbar Extension during Stoop Lifting is Delayed by the Load and Hamstring Tightness. J Phys Ther Sci. 2014 Jan;26(1):57-61. doi: 10.1589/jpts.26.57. Epub 2014 Feb 6. PMID 24567676
- [Background] Houston MN, Hodson VE, Adams KK, Hoch JM. The effectiveness of whole-body-vibration training in improving hamstring flexibility in physically active adults. J Sport Rehabil. 2015 Feb;24(1):77-82. doi: 10.1123/JSR.2013-0059. PMID 25606860
- [Background] Lim KI, Nam HC, Jung KS. Effects on hamstring muscle extensibility, muscle activity, and balance of different stretching techniques. J Phys Ther Sci. 2014 Feb;26(2):209-13. doi: 10.1589/jpts.26.209. Epub 2014 Feb 28. PMID 24648633
- [Background] Michaeli A, Tee JC, Stewart A. DYNAMIC OSCILLATORY STRETCHING EFFICACY ON HAMSTRING EXTENSIBILITY AND STRETCH TOLERANCE: A RANDOMIZED CONTROLLED TRIAL. Int J Sports Phys Ther. 2017 Jun;12(3):305-313. PMID 28593083